CLINICAL TRIAL: NCT03672448
Title: Shanghai Mental Health Center, Shanghai Jiaotong University School of Medicine
Brief Title: The China Longitudinal Aging Study of Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: CRC2017ZD02
Record Dates: First submitted 2018-01-26; First posted 2018-09-14 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Dementia, Vascular; Dementia With Lewy Bodies; Dementia Frontal; Depression; Anxiety
Keywords: dementia; depression; cohort study; sample bank; precision diagnosis; brain imaging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Depression; Anxiety Disorders; Dementia | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and mRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurocognitive disorder: Dementias
  Interventions: Other: Naturalistic observation
- Normal Aging: Normal Aging with normal cognitive function
  Interventions: Other: Naturalistic observation

INTERVENTIONS:
Other: Naturalistic observation — Naturalistic observation
  Other Names: Normal Aging

SUMMARY:
Alzheimer's disease (AD) and Vascular dementia (VaD) have become common diseases in the elderly. The burden of dementia is rising in China, with major medical, social and economic impacts. To address this important public health problem, cohort study on elderly cognitive disorders should be carry out. The methods of early prevention, early diagnosis and early treatment the cognitive disorders in elderly should be found to reduce the burden of the social and economic issue due to dementia. At present, the international corresponding guidelines have taken gene and brain imaging biomarkers as important indicators of dementia pathogenesis research, accurate diagnosis and targeted intervention. Based on the above understanding, the study carry out the population cohort study based on accurate diagnosis and construct the high standard information and sample bank. The study will establish the standard and quality system of geriatric cognitive disorders cohort study (unified standards and norms). The study will integrate the standard biological samples stratified acquisition function module (homogeneity and precision) of elderly cognitive disorders, and complete the construction of biological samples bank and clinical diagnosis and treatment information database. The study will apply and develop brain structural and pathological imaging technology to support precision diagnosis of senile cognitive disorders. The study will evaluate whether peripheral nerve degeneration can predict central nervous system degeneration based on the large cohort of elderly study. In addition, The study will make an effective supplement the sample bank construction of Shanghai Mental Health Center.

DETAILED DESCRIPTION:
The neuropsychological test battery are used to access the cognitive function of subjects in the study. The brain MRI and biochemical examination will be done in the screening period. The samples such as plasma, serum, urine and faeces et al. of the subjects will be collected in the study.

ELIGIBILITY:
Inclusion Criteria:

* registered residents in the community;
* ≥ 60 years;
* without schizophrenia or mental retardation;
* be able to communicate and accept physical and cognitive examinations

Exclusion Criteria:

* blind
* deaf mute

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10,000 adult Chinese aged 60 and up who have been living Shanghai will be recruited.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence, incidence of neurocognitive disorder | 5 years
  Prevalence, incidence of neurocognitive disorder such as AD, MCI and other types of dementia

SECONDARY OUTCOMES:
Prevalence, incidence of mood disorder | 5 years
  Prevalence, incidence of mood disorder such as depression, anxiaty
conversion rate | 5 years
  conversion rate of neurocognitive disorder from Normal Elderly

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Centre
Locations (1):
- Shanghai Mental Health Centre, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang T, He H, Shi Y, Su N, Zhu M, Yan F, Liu Y, Li J, Tang M, Chen W, Bao F, Wang H, Wang Y, Liu Y, Yuan Y, Zuo X, Zhang X, Cui L, Wu W, Zhang C, Lu Y, Fang Y, Xiao S. Prevalence, incidence and modifiable factors for subtypes of mild cognitive impairment: results from the Longitudinal Ageing Study in China. Gen Psychiatr. 2025 Mar 7;38(2):e101736. doi: 10.1136/gpsych-2024-101736. eCollection 2025. PMID 40070969